CLINICAL TRIAL: NCT04211207
Title: Evaluation of the Heart's Respiratory Quotient as Predictive Value After Extra-hospital
Brief Title: Evaluation of the Heart's Respiratory Quotient as Predictive Value After Extra-hospital Cardiac Arrest
Acronym: QUANTIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.296; 2019-A02548-49 (Other: ID RCB)
Record Dates: First submitted 2019-12-17; First posted 2019-12-26 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Arrest
Keywords: Heart's respiratory quotient; Cardiac Arrest; Non-invasive monitoring; Poor prognosis
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non invasive monitoring value — heart's respiratory quotient as non invasive monitoring value

SUMMARY:
It has been shown that elevation of the heart's respiratory quotient after cardiac surgery is predictive of the complications occurrence. In addition, a high heart's respiratory quotient is predictive of anaerobic metabolism after cardiac surgery. In the wake of cardiorespiratory arrest, the presence of anaerobic metabolism reflected by hyperlactatemia is an important prognostic factor. However, this monitoring is invasive and discontinuous. The hypothesis of the study is to show that a rise in the respiratory quotient by a non-invasive monitoring is a factor of poor prognosis in the wake of a Cardiac Arrest.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* Admission to intensive care unit after a non-hospital cardiopulmonary arrest.
* Resumption of spontaneous cardiac activity.
* Non-opposition of the patient or his relatives

Exclusion Criteria:

* Pregnancy
* Prior neurological impairment
* Persons deprived of their liberty by a judicial proceeding, or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ICU for cardiac arrest will be recruited into the study according the inclusion /non inclusion criteria, The patient should be inclued according the investigtor decision, and the non-opposition of patient's relatives was asked as soon as possible. the eligible patient will be enrolled in the study and post cardiac arrest standard care was applied, Implementation of the calorimetry module for the constants collection. data collection was during the first 24 hours.
  When the patient wakes up: information and collection of his non-opposition was asked. The vital status will be collected at 30 day and neurological prognosis evaluation defined by the CPC scorewill be collected at 90 ± 7j by telephone contact.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Heart's respiratory value at H6 post intensive care unit admission to predict mortality | At 6 hours post intensive care unit admission
  Physiological parameter

SECONDARY OUTCOMES:
Heart's respiratory value at intensive care unit admission to predict mortality | At admission of intensive care unit
  Physiological parameter
Heart's respiratory value at H12 post intensive care unit admission to predict mortality | At 12 hours post intensive care unit admission
  Physiological parameter
Heart's respiratory value at H24 post intensive care unit admission to predict mortality | At 24 hours post intensive care unit admission
  Physiological parameter
Heart's respiratory value at intensive care unit admission to predict neurological prognosis | At admission of intensive care unit
  Physiological parameter
Heart's respiratory value at H6 post intensive care unit admission to predict neurological prognosis | At 6 hours post intensive care unit admission
  Physiological parameter
Heart's respiratory value at H12 post intensive care unit admission to predict neurological prognosis | At 12 hours post intensive care unit admission
  Physiological parameter
Heart's respiratory value at H24 post intensive care unit admission to predict neurological prognosis | At 24 hours post intensive care unit admission
  Physiological parameter
metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict mortality at intensive care unit admission | At admission of intensive care unit
  Metabolic parameters
metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict mortality at H6 post intensive care unit admission | At 6 hours post intensive care unit admission
  Metabolic parameters
Metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict mortality at H12 post intensive care unit admission | At 12 hours post intensive care unit admission
  Metabolic parameters
Metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict mortality at H24 post intensive care unit admission | At 24 hours post intensive care unit admission
  Metabolic parameters
Metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict neurological prognosis at intensive care unit admission | At admission of intensive care unit
  Metabolic parameters
Metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict neurological prognosis at H6 post intensive care unit admission | At 6 hours post intensive care unit admission
  Metabolic parameters
Metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict neurological prognosis at H12 post intensive care unit admission | At 12 hours post intensive care unit admission
  Metabolic parameters
Metabolic parameters ( lactate, Oxygen consummation, carbon dioxide production and central venous oxygen saturation) to predict neurological prognosis at H24 post intensive care unit admission | At 24 hours post intensive care unit admission
  Metabolic parameters
Cardiac arrest circumstances following Utstein-style guidelines according mortality | At admission of intensive care unit
  Metabolic parameters
Cardiac arrest circumstances following Utstein-style guidelines according neurological prognosis | At admission of intensive care unit
  Cardiac arrest circumstances
Vital status at day 30 | At 30 Days post intensive car unit admission
  Alive or Dead status
Cerebral performance category (CPC) score at day 90 | At 90 Days post intensive car unit admission
  Cerebral performance category (CPC) score : CPC=1 : Conscious, alert, and oriented with normal cognitive functions, CPC=2 : Conscious and alert with moderate cerebral disability; CPC=3: Conscious with severe disability; CPC=4: Comatose or in persistent vegetative state; CPC=5 : Certified brain death or dead by traditional criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luc G, Baert V, Escutnaire J, Genin M, Vilhelm C, Di Pompeo C, Khoury CE, Segal N, Wiel E, Adnet F, Tazarourte K, Gueugniaud PY, Hubert H; On behalf GR-ReAC. Epidemiology of out-of-hospital cardiac arrest: A French national incidence and mid-term survival rate study. Anaesth Crit Care Pain Med. 2019 Apr;38(2):131-135. doi: 10.1016/j.accpm.2018.04.006. Epub 2018 Apr 21. PMID 29684654
- [Background] Horburger D, Testori C, Sterz F, Herkner H, Krizanac D, Uray T, Schober A, Stockl M, Stratil P, Weiser C, Wallmuller C, Holzer M. Mild therapeutic hypothermia improves outcomes compared with normothermia in cardiac-arrest patients--a retrospective chart review. Crit Care Med. 2012 Aug;40(8):2315-9. doi: 10.1097/CCM.0b013e31825333cf. PMID 22622403
- [Background] Bhattacharjee S, Baidya DK, Maitra S. Therapeutic hypothermia after cardiac arrest is not associated with favorable neurological outcome: a meta-analysis. J Clin Anesth. 2016 Sep;33:225-32. doi: 10.1016/j.jclinane.2016.03.001. Epub 2016 May 5. PMID 27555170
- [Background] Adnet F, Triba MN, Borron SW, Lapostolle F, Hubert H, Gueugniaud PY, Escutnaire J, Guenin A, Hoogvorst A, Marbeuf-Gueye C, Reuter PG, Javaud N, Vicaut E, Chevret S. Cardiopulmonary resuscitation duration and survival in out-of-hospital cardiac arrest patients. Resuscitation. 2017 Feb;111:74-81. doi: 10.1016/j.resuscitation.2016.11.024. Epub 2016 Dec 14. PMID 27987396
- [Background] Lemiale V, Dumas F, Mongardon N, Giovanetti O, Charpentier J, Chiche JD, Carli P, Mira JP, Nolan J, Cariou A. Intensive care unit mortality after cardiac arrest: the relative contribution of shock and brain injury in a large cohort. Intensive Care Med. 2013 Nov;39(11):1972-80. doi: 10.1007/s00134-013-3043-4. Epub 2013 Aug 14. PMID 23942856
- [Background] Pekkarinen PT, Backlund M, Efendijev I, Raj R, Folger D, Litonius E, Laitio R, Bendel S, Hoppu S, Ala-Kokko T, Reinikainen M, Skrifvars MB. Association of extracerebral organ failure with 1-year survival and healthcare-associated costs after cardiac arrest: an observational database study. Crit Care. 2019 Feb 28;23(1):67. doi: 10.1186/s13054-019-2359-z. PMID 30819234
- [Background] Dell'Anna AM, Sandroni C, Lamanna I, Belloni I, Donadello K, Creteur J, Vincent JL, Taccone FS. Prognostic implications of blood lactate concentrations after cardiac arrest: a retrospective study. Ann Intensive Care. 2017 Oct 6;7(1):101. doi: 10.1186/s13613-017-0321-2. PMID 28986863
- [Background] Kliegel A, Losert H, Sterz F, Holzer M, Zeiner A, Havel C, Laggner AN. Serial lactate determinations for prediction of outcome after cardiac arrest. Medicine (Baltimore). 2004 Sep;83(5):274-279. doi: 10.1097/01.md.0000141098.46118.4c. PMID 15342971
- [Background] Riveiro DF, Oliveira VM, Braunner JS, Vieira SR. Evaluation of Serum Lactate, Central Venous Saturation, and Venous-Arterial Carbon Dioxide Difference in the Prediction of Mortality in Postcardiac Arrest Syndrome. J Intensive Care Med. 2016 Sep;31(8):544-52. doi: 10.1177/0885066615592865. Epub 2015 Jun 24. PMID 26112759
- [Background] Cocchi MN, Miller J, Hunziker S, Carney E, Salciccioli J, Farris S, Joyce N, Zimetbaum P, Howell MD, Donnino MW. The association of lactate and vasopressor need for mortality prediction in survivors of cardiac arrest. Minerva Anestesiol. 2011 Nov;77(11):1063-71. Epub 2011 May 11. PMID 21597442
- [Background] Walley KR. Use of central venous oxygen saturation to guide therapy. Am J Respir Crit Care Med. 2011 Sep 1;184(5):514-20. doi: 10.1164/rccm.201010-1584CI. PMID 21177882
- [Background] Rivers EP, Rady MY, Martin GB, Fenn NM, Smithline HA, Alexander ME, Nowak RM. Venous hyperoxia after cardiac arrest. Characterization of a defect in systemic oxygen utilization. Chest. 1992 Dec;102(6):1787-93. doi: 10.1378/chest.102.6.1787. PMID 1446489
- [Background] Gaieski DF, Band RA, Abella BS, Neumar RW, Fuchs BD, Kolansky DM, Merchant RM, Carr BG, Becker LB, Maguire C, Klair A, Hylton J, Goyal M. Early goal-directed hemodynamic optimization combined with therapeutic hypothermia in comatose survivors of out-of-hospital cardiac arrest. Resuscitation. 2009 Apr;80(4):418-24. doi: 10.1016/j.resuscitation.2008.12.015. Epub 2009 Feb 12. PMID 19217200
- [Background] Walters EL, Morawski K, Dorotta I, Ramsingh D, Lumen K, Bland D, Clem K, Nguyen HB. Implementation of a post-cardiac arrest care bundle including therapeutic hypothermia and hemodynamic optimization in comatose patients with return of spontaneous circulation after out-of-hospital cardiac arrest: a feasibility study. Shock. 2011 Apr;35(4):360-6. doi: 10.1097/SHK.0b013e318204c106. PMID 21068697
- [Background] Mallat J, Lemyze M, Tronchon L, Vallet B, Thevenin D. Use of venous-to-arterial carbon dioxide tension difference to guide resuscitation therapy in septic shock. World J Crit Care Med. 2016 Feb 4;5(1):47-56. doi: 10.5492/wjccm.v5.i1.47. eCollection 2016 Feb 4. PMID 26855893
- [Background] Solberg G, Robstad B, Skjonsberg OH, Borchsenius F. Respiratory gas exchange indices for estimating the anaerobic threshold. J Sports Sci Med. 2005 Mar 1;4(1):29-36. eCollection 2005 Mar 1. PMID 24431958
- [Background] Mekontso-Dessap A, Castelain V, Anguel N, Bahloul M, Schauvliege F, Richard C, Teboul JL. Combination of venoarterial PCO2 difference with arteriovenous O2 content difference to detect anaerobic metabolism in patients. Intensive Care Med. 2002 Mar;28(3):272-7. doi: 10.1007/s00134-002-1215-8. Epub 2002 Feb 8. PMID 11904655
- [Background] Mukai A, Suehiro K, Kimura A, Funai Y, Matsuura T, Tanaka K, Yamada T, Mori T, Nishikawa K. Comparison of the venous-arterial CO2 to arterial-venous O2 content difference ratio with the venous-arterial CO2 gradient for the predictability of adverse outcomes after cardiac surgery. J Clin Monit Comput. 2020 Feb;34(1):41-53. doi: 10.1007/s10877-019-00286-z. Epub 2019 Feb 22. PMID 30796642
- [Background] Piot J, Hebrard A, Durand M, Payen JF, Albaladejo P. An elevated respiratory quotient predicts complications after cardiac surgery under extracorporeal circulation: an observational pilot study. J Clin Monit Comput. 2019 Feb;33(1):145-153. doi: 10.1007/s10877-018-0137-0. Epub 2018 Apr 17. PMID 29667097
- [Background] Shinozaki K, Becker LB, Saeki K, Kim J, Yin T, Da T, Lampe JW. Dissociated Oxygen Consumption and Carbon Dioxide Production in the Post-Cardiac Arrest Rat: A Novel Metabolic Phenotype. J Am Heart Assoc. 2018 Jun 29;7(13):e007721. doi: 10.1161/JAHA.117.007721. PMID 29959138
- [Background] Uber A, Grossestreuer AV, Ross CE, Patel PV, Trehan A, Donnino MW, Berg KM. Preliminary observations in systemic oxygen consumption during targeted temperature management after cardiac arrest. Resuscitation. 2018 Jun;127:89-94. doi: 10.1016/j.resuscitation.2018.04.001. Epub 2018 Apr 4. PMID 29626611